CLINICAL TRIAL: NCT07023380
Title: Pilot Interventional Study of an EoE-Causal Food Identification Blood Test
Brief Title: EoE Food Test Pilot Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Food Allergy Fund (Unknown); American Partnership for Eosinophilic Disorders (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24-022349
Record Dates: First submitted 2025-06-10; First posted 2025-06-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Eosinophilic Esophagitis Caused by Food (Disorder)

STUDY DESIGN:
Intervention Model Description: This pilot interventional prospective cohort study will enroll subjects with Eosinophilic esophagitis (EoE) who have not yet identified causal foods. Subject blood will be drawn and food-activated T cell responses will be assayed. Test results will be provided to subjects physician(s) to be used in conjunction with standard-of-care practices when determining which foods should be removed from the subject's diet. Symptoms and inflammation will be measured by PEESS Child and Parent Surveys and standard of care (SOC) endoscopy with esophageal biopsy, respectively. Response to research assay-aided diet changes will provide information about the assay's clinical value in a "real-world" setting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EoE unknown (Experimental): Patients with Eosinophilic esophagitis who have not yet identified their disease causal foods and are interested in an elimination diet approach to disease management
  Interventions: Diagnostic Test: Assay directed diet change

INTERVENTIONS:
Diagnostic Test: Assay directed diet change — Functional T cell assay(s) will be performed on research subjects' peripheral blood using four foods known to commonly cause Eosinophilic esophagitis - milk, soy, egg, and wheat. Response magnitude to foods in vitro will influence whether a subject's physician chooses to recommend the subject AVOID the food or continue to CONSUME the food. Disease response to the diet changes will be evaluated in standard-of-care follow up endoscopy.

SUMMARY:
The objective of this study is to determine the performance characteristics of a series of novel, non-invasive allergen-activated T cell assays designed to identify Eosinophilic esophagitis (EoE) causal foods, when used in conjunction with standard-of-care (SOC) practices.

The question it aims to answer is:

Will assay results accurately predict EoE food allergies in concordance with SOC endoscopies after diet changes?

DETAILED DESCRIPTION:
This proof-of-concept, interventional prospective cohort study will enroll subjects with Eosinophilic esophagitis (EoE) who have not yet identified causal foods. Subject blood will be drawn and food-activated T cell responses will be assayed. Subjects will be advised to remove foods based on standard-of-care practices and/or the outcome of their T cell assays ("personalized elimination diet"). Symptoms will be measured by the Pediatric Eosinophilic Esophagitis Symptom Scores (PEESS) Child and Parent Surveys and standard of care (SOC) endoscopy with esophageal biopsy, respectively. Response to research assay-directed diet changes will provide information about the assay's clinical value.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of Eosinophilic esophagitis (EoE) based on positive esophageal biopsy (>15 eosinophils/high power field) within three months of enrollment.

AND Intention to undergo dietary intervention for treatment of their EoE. AND Unknown contribution of one or more of milk, soy, egg, and wheat to their EoE disease state.

AND Willingness to adopt an elimination diet based in part on the results of the experimental testing.

Exclusion Criteria:

Proton pump inhibitor (PPI)-responsive EoE: Resolution or response of EoE to high-dose PPI (2 mg/kg) alone, at the PI's discretion.

OR Presence of other inflammatory or infectious gastrointestinal pathology (e.g. eosinophilic gastrointestinal diseases, irritable bowel disease, Infectious Colitis, etc.), at the discretion of the Principal Investigator (PI).

OR Prior medical or surgical history that precludes safely performing an upper endoscopy with biopsy or restriction of diet.

OR Current immunomodulatory therapy >4 weeks (swallowed or systemic steroids, biologic therapy, chemotherapy. etc.) that may interfere with the blood test or biopsy results, at the PI's discretion.

OR Inability to read or understand English.

Ages: 0 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Esophageal eosinophilia (number of eosinophils in the esophagus) | At least 4 weeks after implementation of diet changes
  Eosinophils per high power field on follow up esophageal biopsy

SECONDARY OUTCOMES:
Pediatric Eosinophilic Esophagitis Symptom Score (total score based on pediatric symptom score) | At least 4 weeks after implementation of diet changes
  Min 0-Max 100 (lower is better)

CONTACTS AND LOCATIONS:
Overall Officials: David A Hill, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia, University of Pennsylvania
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data with other researchers. All data that may be published or shared with other researchers will be deidentified and will not include information such as informed consent forms.

REFERENCES:
- [Background] Hill DA, Spergel JM. The Immunologic Mechanisms of Eosinophilic Esophagitis. Curr Allergy Asthma Rep. 2016 Feb;16(2):9. doi: 10.1007/s11882-015-0592-3. PMID 26758862
- [Background] De Vlieger L, Smolders L, Nuyttens L, Verelst S, Breynaert C, Vanuytsel T, Hoffman I, Bullens DM. A Clinical Perspective on the Dietary Therapies for Pediatric Eosinophilic Esophagitis: The Gap Between Research and Daily Practice. Front Immunol. 2021 May 19;12:677859. doi: 10.3389/fimmu.2021.677859. eCollection 2021. PMID 34093578
- [Background] Nhu QM, Aceves SS. Tissue Remodeling in Chronic Eosinophilic Esophageal Inflammation: Parallels in Asthma and Therapeutic Perspectives. Front Med (Lausanne). 2017 Aug 7;4:128. doi: 10.3389/fmed.2017.00128. eCollection 2017. PMID 28831387
- [Background] Spergel JM, Brown-Whitehorn TF, Cianferoni A, Shuker M, Wang ML, Verma R, Liacouras CA. Identification of causative foods in children with eosinophilic esophagitis treated with an elimination diet. J Allergy Clin Immunol. 2012 Aug;130(2):461-7.e5. doi: 10.1016/j.jaci.2012.05.021. Epub 2012 Jun 27. PMID 22743304
- [Background] Dellon ES, Rusin S, Gebhart JH, Covey S, Higgins LL, Beitia R, Speck O, Woodward K, Woosley JT, Shaheen NJ. Utility of a Noninvasive Serum Biomarker Panel for Diagnosis and Monitoring of Eosinophilic Esophagitis: A Prospective Study. Am J Gastroenterol. 2015 Jun;110(6):821-7. doi: 10.1038/ajg.2015.57. Epub 2015 Mar 17. PMID 25781367
- [Background] Dilollo J, Rodriguez-Lopez EM, Wilkey L, Martin EK, Spergel JM, Hill DA. Peripheral markers of allergen-specific immune activation predict clinical allergy in eosinophilic esophagitis. Allergy. 2021 Nov;76(11):3470-3478. doi: 10.1111/all.14854. Epub 2021 May 14. PMID 33840099